CLINICAL TRIAL: NCT06735573
Title: Observational Study to Explore the Relationship Between Dietary Protein Intake and the Prevalence of Sarcopenic Obesity in Adult Female With Chronic Obstructive Pulmonary Disease (COPD): A Pilot Study
Brief Title: Protein, Sarcopenic Obesity, and COPD
Acronym: PROSO-COPD
Status: Not yet recruiting | Type: Observational
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Other Study IDs: T Baabbad; University of Aberdeen (Other: University of Aberdeen)
Record Dates: First submitted 2024-12-05; First posted 2024-12-16 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Sarcopenic Obesity; Chronic Obstructive Pulmonary Diseases
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — A single blood sample will be taken by venepuncture (usually from the antecubital vein) by a trained phlebotomist, after at least 9 hours of fasting overnight. The blood sample will be collected into a heparin tube and spun (for 15 minutes at 2000 x g) to obtain plasma. Plasma samples will be stored at - 80°C until batch analysis of high-sensitivity C-reactive protein (hs-CRP) levels, using the Konelab Clinical Analyser at the Rowett Institute, the University of Aberdeen, Aberdeen, United Kingdom.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: the relationship between the quantity and source of dietary protein intake, and the prevalence of sarcopenic obesity, and lung function outcomes — Primary Objective The primary objective is to measure the relationship between the quantity and source of dietary protein intake, and the prevalence of sarcopenic obesity, and lung function outcomes, in older female participants with clinically diagnosed COPD.
  Secondary Objectives The secondary objective is to investigate whether the level of inflammation (plasma CRP) is associated with the intake of total, plant-based and animal-based protein, with the prevalence of sarcopenic obesity, and with lung function outcomes.
  Other Names: the level of inflammation (plasma CRP)

SUMMARY:
Both sarcopenic obesity and chronic obstructive pulmonary diseases (COPD) are common conditions that mainly affect middle-aged and older adults. Previous research has shown that increased dietary intake of total and plant-based protein is associated with a lower risk of sarcopenic obesity, using data from the EPIC Norfolk study. Furthermore, a systematic review and meta-analysis showed that having sarcopenic obesity was associated with significantly impaired lung function outcomes. Other research has shown that increased intake of dietary protein leads to a better treatment outcome for respiratory diseases. The aim of this pilot observational study is to investigate, in more detail, the relationship between the quantity and source of dietary protein intake, the prevalence of sarcopenic obesity, and lung function, in a small cohort of older female participants with COPD. The study will also consider the role of inflammation in relation to sarcopenic obesity and lung function outcomes. This study will help to improve the understanding of the relationship between sarcopenic obesity and lung function outcomes, and how dietary protein intake and inflammation can affect this relationship and each of the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Women.
* Clinically diagnosed with COPD.
* Aged 55 years or older.

Exclusion Criteria:

* Male.
* Women who are 54 years or younger.
* Those who have dementia.
* Unable to read or write in English.
* Unable to attend the Human Intervention Studies Unit.
* Those within one year life expectancy.
* Those who have cancer.

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female with COPD aged 55 and over
Study Population: Women with clinically diagnosed COPD, from GP practices in Aberdeen,United Kingdom, through the Primary Care Research Network.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Association between dietary protein and the prevalence of sarcopenic obesity | through study completion, an average of 1 year
  Association between dietary intake of total, plant-based and animal-based protein and the prevalence of sarcopenic obesity.

SECONDARY OUTCOMES:
Association between dietary protein and lung functions outcomes | through study completion, an average of 1 year
  Association between dietary intake of total, plant-based and animal-based protein and lung functions outcomes (Forced Vital Capacity (FVC), Forced Expiratory Volume in The First Second(FEV1), and The Ratio of Forced Expiratory Volume in The First Second to Forced Vital Capacity (FEV1/FVC ratio)).

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.